CLINICAL TRIAL: NCT04464889
Title: A Dose-Escalation, Open Label Phase I Study to Assess the Safety, Feasibility and Preliminary Efficacy of HA-1H TCR Modified T Cells, MDG1021, in Patients With Relapsed or Persistent Hematologic Malignancies After Allogeneic HSCT With or Without Unmanipulated DLI
Brief Title: HA-1H TCR T Cell for Relapsed/Persistent Hematologic Malignancies After Allogeneic Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Medigene transfered all rights to a new Sponsor
Sponsor: Medigene AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-TCR-003
Record Dates: First submitted 2020-07-01; First posted 2020-07-09 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Disorders; Chronic Myeloid Leukemia; Myelofibrosis; Multiple Myeloma; Malignant Lymphoma
Keywords: Allogeneic hematopoietic stem cell transplantation; Relapsed hematologic malignancy; Persistent hematologic malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis; Multiple Myeloma; Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: The aim of the study is to determine the recommended phase II dose (RP2D) of MDG1021 that will be determined on the basis of safety and ability to manufacture a cohort specific MDG1021 dose. The dose-escalation part of the study is designed to assess the safety and the MTD of MDG1021, using a standard 3+3 cohort design, with up to 3 additional subjects to be enrolled in case of dose limiting toxicity (DLT).
  Upon completion of the dose-escalation part of the study, 20 eligible patients will be treated in the expansion part of the study with MDG1021 at the RP2D to further evaluate safety, feasibility and preliminary efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDG1021 (Experimental): Dose-escalation part of the study to investigate 3 MDG1021 doses. Dose-expansion part of the study to investigate the selected optimal MDG1021 dose.
  Interventions: Drug: MDG1021 dose 1; Drug: MDG1021 dose 2; Drug: MDG1021 dose 3; Drug: MDG1021 optimal dose

INTERVENTIONS:
Drug: MDG1021 dose 1 — 3 patients to receive dose1: target dose of 0.3x10^6 HA-1H TCR transduced T cells/kg BW ±20% in 100 mL
Drug: MDG1021 dose 2 — 3 patients to receive dose 2: target dose of 1x10^6 HA-1H TCR transduced T cells/kg BW ±20% in 100 mL
Drug: MDG1021 dose 3 — 3 patients to receive dose 3: target dose of 3x10^6 HA-1H TCR transduced T cells/kg BW +20% in 100 mL
Drug: MDG1021 optimal dose — 20 patients to receive the selected optimal dose

SUMMARY:
This is a non-randomised, open-label phase I study of an investigational medicinal product (IMP) consisting of a HLA-A*02:01 restricted HA-1H T cell receptor transduced T cell (MDG1021) immunotherapy for relapsed or persistent hematologic malignancies after allogeneic hematopoietic stem cell transplantation. The aim of the study is to determine the recommended phase II dose of MDG1021.

DETAILED DESCRIPTION:
This phase I is designed to assess the safety and feasibility of a HLA-A*02:01 restricted, HA-1H T cell receptor (TCR) transduced patient-derived T cell (MDG1021) immunotherapy, with secondary endpoints including preliminary efficacy, in patients with relapsed or persistent hematologic malignancies after allogeneic hematopoietic stem cell transplantation. In the dose-escalation part of the study, at least 9 patients will be treated with MDG1021 at 3 different doses to assess the safety and the maximum tolerated dose using a standard 3+3 cohort design. Thereafter, the selected optimal MDG1021 dose will be assessed for safety and preliminary efficacy in 20 additional patients during the dose-expansion part of the study. Manufacturing feasibility will be determined. MDG1021 will be administered by single intravenous infusion.

HA-1H is exclusively expressed on cells of the hematopoietic system. If the patient's blood-cells, and thus lymphoma or leukemic cells, carry the immunogenic version of the HA-1H antigen on their surface and the donor stem cells do not, MDG1021 immunotherapy could eradicate the patient's cancer cells and allow the donor stem cells to repopulate the patient's blood forming system.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or persistent disease is defined according to disease specific guidelines (AML, CML, MM, ALL, MDS, MPN, MF and malignant B- or T-cell lymphoma) and includes MRD positivity.
2. Patients positive for HLA-A*02:01 according to genotyping results
3. Patients positive for HA-1H
4. Patients who received the allo-HSCT at least 100 days preceding the leukapheresis
5. Patients (i.e. recipient) transplanted with a sibling or unrelated HSCT donor

   1. donor being HLA-A*02:01 positive and HA-1H negative, or
   2. a donor with a single mismatch at HLA-A*02:01, being HA-1H positive or negative
6. Patients from whom at least 10x10^6 donor CD8+ T cells can be harvested by leukapheresis
7. Age ≥ 18 years, of either sex
8. ECOG performance status 0-2.
9. Life expectancy of at least 3 months
10. Patients must be able to understand and be willing to give signed informed consent

Exclusion Criteria:

1. Evidence of acute or chronic graft versus host disease (GVHD) ≥ grade II
2. Serologic evidence of acute or chronic hepatitis B virus infection (i.e. positive for HBsAg or IgM anti-HBc). Positive HIV and HCV serology or active bacterial infection
3. Medical or psychological conditions that would make the patient unsuitable candidate for cell therapy at the discretion of the investigator. Special risks to be considered:

   1. Creatinine > 2.5 times the upper limit of normal (ULN) serum level
   2. Total bilirubin, ALAT, ASAT > 3.0 x ULN serum level
   3. Cardiac left ventricular ejection fraction < 35% at rest
   4. Severe restrictive or obstructive lung disease
4. Clinically significant and ongoing immune suppression including, but not limited to immunosuppressive agents (e.g. cyclosporine or corticosteroids (at an equivalent dose of ≥ 10 mg prednisone per day)). Inhaled steroid and physiological replacement for adrenal insufficiency is allowed
5. Patients with a history of primary immunodeficiency
6. Patients with a currently active second malignancy other than nonmelanoma skin cancers or subjects with history of prior malignancy and previously treated with a curative intent therapy less than 1 year ago
7. Patients both with urinary outflow obstructions and on dialysis or patients for whom cyclophosphamide is contraindicated for other reasons
8. Known or suspected hypersensitivity or intolerance to IMP, cyclophosphamide, fludarabine and/or tocilizumab or to any of the excipients
9. Participation in any clinical study < 60 days prior to first IMP administration in case of antibodies and < 14 days for all other IMPs
10. Vulnerable patients and/or patients unwilling or unable to comply with procedures required in this clinical study protocol
11. Pregnant or lactating women
12. Women of child-bearing potential not using highly effective method(s) of birth control (i.e., with low failure rate < 1% per year) throughout the study and/or unwilling to be tested for pregnancy. A negative serum β-hCG test is required at baseline
13. Fertile men not agreeing to use effective contraceptive methods during the clinical study

    Exclusion criteria at time of IMP administration:
14. Uncontrolled central nervous system (CNS) disease
15. Uncontrolled, life threatening infections or uncontrolled disseminated intravascular coagulation; however, if these problems resolve, the start of treatment can be initiated on a delayed schedule
16. Evidence of acute or chronic graft versus host disease (GVHD) ≥ grade II
17. Unable to generate HA-1H TCR transduced T cells for transfusion (out of specification). However, if a lower than planned number of cells is available, the patient will have the option to receive the OOS HA-1H TCR transduced T cells product (cell dose must be at least the lowest dose level of D1 and will be analyzed in the safety and full analysis set populations.
18. If not enough starting material is collected during leukapheresis, the patient will be excluded from study participation and receive best available standard therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of HA-1H TCR transduced T cells: incidence and severity of adverse events | up to 28 days after T cell infusion
  To assess the incidence and severity of adverse events during the dose escalation part of the study according to the NCI CTCAE v5.0
Maximum tolerated dose (MTD) of HA-1H TCR transduced T cells | up to 28 days after T cell infusion
  To asses the maximum tolerated dose (MTD) of MDG1021 as determined by dose-limiting toxicities (DLTs)
Recommended phase 2 dose (RP2D) of HA-1H TCR transduced T cells | up to 28 days after T cell infusion
  To asses the recommended phase II dose (RP2D) of MDG1021
Safety and tolerability of HA-1H TCR transduced T cells at recommended phase II dose: incidence and severity of adverse events | up to 28 days after T cell infusion
  To assess the incidence and severity of adverse events of MDG1021 at the RP2D during the expansion part of the study according to the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Safety and tolerability (both parts of the study): incidence and severity of adverse events | Up to 12 months after T cell infusion
  To assess the incidence and severity of AEs ≥ grade 3 (NCI CTCAE v5.0)
Overall response rate | Up to 12 months after T cell infusion
  To assess the overall response rate defined as the proportion of patients with a best overall response of complete response (CR), partial response (PR), and/or their disease specific subcategories
Overall survival | Up to 12 months afterT cell infusion
  To assess the overall survival (OS) defined as the time from the date of signing the informed consent until the documented date of death.
Progression free survival | Up to 12 months afterT cell infusion
  To assess the progression-free survival (PFS) defined as the time from the date of signing the date of signed informed consent until progressive disease/relapse or death, whichever occurs first.
Duration of response | Up to 12 months afterT cell infusion
  To assess the duration of response (DoR) defined as time from the date of the first documented response to the first documented progression of disease or death due to underlying cancer.
Quality of life (EQ-5D-5L) | Up to 12 months afterT cell infusion
  The quality of life will be assessed by using the EQ-5D-5L questionnaire, consisting of 5 questions. Higher scores correspond to higher quality of life.
Quality of life (VAS) | Up to 12 months afterT cell infusion
  The quality of life will be assessed by a visual analog scale (EuroQoL), having a range of 0 ot 100, with higher scores corresponding to better quality of life.

OTHER OUTCOMES:
Feasibility of manufacturing HA-1H TCR transducer T cells: proportion of patients for whom leukapheresis was feasible | Up to Day 0 after T cell infusion
  Feasibility is determined by the proportion of patients for whom leukapheresis was feasible, for whom manufacturing MDG1021 was feasible, and whom received MDG1021 by intravenous infusion
Persistence and expansion of HA-1H transduced T cells in peripheral blood | Up to 12 months afterT cell infusion
  To evaluate the persistence (flow cytometry with tetramers evaluating the % HA-1H transduced T cells among all T cells) and expansion of HA-1H transduced T cells (as % HA-1H transduced T cells among all T cells over time) in peripheral blood
Function of HA-1H TCR transduced T cells detectable in peripheral blood | Up to 12 months afterT cell infusion
  To evaluate the function of HA-1H TCR transduced T cells detectable in peripheral blood by ELISA, measuring Interferon gamma production
Phenotype of HA-1H TCR transduced T cells detectable in peripheral blood | Up to 12 months afterT cell infusion
  To evaluate the phenotype of HA-1H TCR transduced T cells detectable in peripheral blood by flow cytometry of T cell subtypes expressed in % of all T cells
Disappearance of recipient hematopoiesis (chimerism analysis) in the blood | Up to 12 months after T cell infusion
  To evaluate disappearance of recipient hematopoiesis (chimerism analysis) in the blood
Disappearance of recipient hematopoiesis (chimerism analysis) in the bone marrow | Up to 3 months after T cell infusion
  To evaluate disappearance of recipient hematopoiesis (chimerism analysis) in the bone marrow
Other explorative endpoints | Up to 12 months after T infusion
  To investigate biomarkers and molecular signatures, potentially related to safety, anti-tumor activity, the mode-of-action of MDG1021 and the pathophysiology of disease

CONTACTS AND LOCATIONS:
Overall Officials: Peter van Balen, MD, Principal Investigator — Leiden University Medical Centre; Rene Goedkoop, MD, Study Director — Medigene AG
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No